CLINICAL TRIAL: NCT06641544
Title: The Efficacy and Safety of Different Combination Regimens of Inetetamab in First-line Treatment of HER2 Positive Metastatic Breast Cancer
Acronym: IFANS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jianli Zhao, Associate Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SSKY-012
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Group (Active Comparator): Inetetamab：was administered as an intravenous (IV) loading dose of 8mg/kg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 6mg/kg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Pertuzumab：was administered as an intravenous (IV) loading dose of 840mg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 420mg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Chemotherapy regimen chosen by the physician
  Interventions: Drug: Inetetamab
- B Group (Experimental): Inetetamab：was administered as an intravenous (IV) loading dose of 8mg/kg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 6mg/kg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Pyrotinib：400 mg once daily orally within 30 minutes after a meal at the same time each day.
  Chemotherapy regimen chosen by the physician
  Interventions: Drug: Inetetamab

INTERVENTIONS:
Drug: Inetetamab — Group A received Inetetamab+Pertuzumab+TPC, while Group B received Inetetamab+Pyrotinib+TPC.
  Other Names: Pertuzumab，Pyrotinib

SUMMARY:
This study is to explore the efficacy and safety of the first-line treatment of HER2 positive recurrent/metastatic breast cancer with Inetetamab combined with Pertuzumab or Pyrotinib combined with chemotherapy, hoping to have better clinical benefits and provide a new treatment mode for targeted treatment.

DETAILED DESCRIPTION:
In terms of the anti-HER2 mechanism, the binding sites of Inetetamab and Trastuzumab are located in the extracellular domain IV, while the binding site of Pertuzumab is located in the conserved domain II, inhibiting HER2 phosphorylation and blocking downstream signaling pathways. The binding site of Pyrotinib is located in the intracellular tyrosinase active domain, which competes with ATP to block HER2 autophosphorylation and activation. Inetetamab combined with Pertuzumab "dual target" blocks HER2 dimer formation, while Inetetamab combined with Pyrotinib "dual target" inhibition can produce synergistic enhancement of anti-HER2 effect. This study is to explore the efficacy and safety of the first-line treatment of HER2 positive recurrent/metastatic breast cancer with Inetetamab combined with Pertuzumab or Pyrotinib combined with chemotherapy, hoping to have better clinical benefits and provide a new treatment mode for targeted treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years and ≤ 70 years old;
* Pathological diagnosis of HER-2 was positive (definition: immunohistochemical results were + + + or in situ hybridization results were positive);
* Invasive breast cancer confirmed by pathological examination, with evidence of local recurrence or imaging metastasis, and those with local recurrence must be confirmed by the researcher as unable to undergo radical surgery;
* Have not received first-line anti-HER2 treatment or (new) adjuvant anti-HER2 drug treatment that is effective and has been discontinued for more than 12 months;
* ECOG PS score 0-2, expected survival period ≥ 6 months, and able to follow up;
* According to the Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1, there must be at least one clearly measurable and/or assessable lesion present, and the lesion diameter evaluated by CT or MRI must be ≥ 1cm;
* In the absence of blood transfusion or pharmacological treatment (granulocyte colony-stimulating factor/erythropoietin (EPO)/interleukin-11, etc.) within 14 days prior to the first treatment, and organ function must meet the following requirements: absolute neutrophil count (ANC) ≥ 1.5×10^9/L; platelets (PLT) ≥ 90×10^9/L; hemoglobin (Hb) ≥ 90g/L. Blood biochemistry: total bilirubin (TBIL) ≤1.5×ULN,known as Gilbert syndrome patients, TBIL ≤ 2 × ULN; ALT and AST ≤2.5×ULN; and liver metastasis patients require ALT and AST ≤5×ULN; Alkaline phosphatase ≤ 2.5 × ULN; BUN and Cr ≤1.5×ULN;
* Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal, unless drugs known to alter INR and APTT are used;
* Left ventricular ejection fraction (LVEF) ≥50%;
* 12 lead electrocardiogram: Fridericia corrected QT interval (QTcF)<470msec;
* No history of major organs such as the heart, lungs, liver, kidneys, or endocrine system;
* Female patients of childbearing age who have negative pregnancy tests and voluntarily adopt effective and reliable contraceptive measures;
* Voluntarily join this study, sign an informed consent form, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

* Have received other clinical study drugs within 4 weeks prior to the first study drug administration;
* Have received any systematic anti-tumor treatment during the recurrence/metastasis stage (excluding endocrine therapy previously performed for recurrence/metastasis stage);
* During the (new) adjuvant phase, other anti-HER2 treatments were received in addition to trastuzumab, pertuzumab, and pyrotinib;
* Patients who experience disease progression during (new) adjuvant trastuzumab treatment, as well as patients who experience recurrence/metastasis within 12 months after completing (new) adjuvant system treatment;
* Evidence of symptomatic central nervous system metastasis or leptomeningeal disease (patients with brain metastases who have received radiation therapy and have been stable for ≥ 4 weeks can be enrolled);
* Patients with only bone or skin as the sole target lesion;
* Serious heart disease or discomfort, including but not limited to the following situations:

  1. History of heart failure or systolic dysfunction (LVEF<50%);
  2. High risk or treatable angina pectoris or arrhythmia (such as second degree type 2 atrioventricular block or third degree atrioventricular block, ventricular tachycardia);
  3. Clinically significant heart valve disease;
  4. Electrocardiogram indicates transmural myocardial infarction;
  5. Uncontrolled hypertension (excluding stable cases where systolic blood pressure>150 mmHg and/or diastolic blood pressure>90 mmHg can be controlled after stable treatment);
* Gastrointestinal dysfunction or gastrointestinal diseases (including active ulcers);
* Presence of active hepatitis B (HBsAg positive and HBV DNA ≥ 500 IU/mL), hepatitis C (hepatitis C antibody positive and HCV RNA above the upper limit of normal range), and cirrhosis;
* History of immunodeficiency, including HIV infection, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
* There is a third fluid accumulation (such as pleural effusion or ascites) that cannot be controlled by drainage or other methods;
* Suffering from serious accompanying diseases or other comorbidities that may interfere with the planned treatment, or any other circumstances that are not suitable for participation in this study, such as pulmonary infections that require treatment;
* Other malignant tumors within the past five years, except for those cured of cervical, basal cell carcinoma, and squamous cell carcinoma;
* The patient has undergone major surgical procedures or significant trauma within the first 4 weeks of randomization, or is expected to undergo major surgical treatment;
* Peripheral neuropathy of grade ≥ 3 judged according to CTCAE 5.0 standards;
* Those who are known to have a history of allergies to the components of this drug regimen;
* Researchers determine that individuals are not suitable for receiving systemic chemotherapy;
* Pregnant or lactating female patients who are unable to use effective contraception throughout the entire trial period and are of childbearing age;
* The researchers believe that it is not appropriate to participate in this trial, as any other medical, social, or psychological factors may affect safety or compliance with research procedures.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-17 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Tumor assessments every 6 weeks from Baseline until radiographical progressive disease (PD), death (whichever occurred first), up to the primary completion date (up to 2 years)
  An objective response was defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR) determined by investigator using RECIST v1.1 on two consecutive occasions ≥4 weeks apart

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Tumor assessments every 6 weeks from randomization to radiographical PD or death from any cause, whichever occurred first，up to the primary completion date (up to 2 years)
  PFS was defined as the time from first dose to first documented radiographical progressive disease (PD) using RECIST version 1.1, or death from any cause , whichever occurred first.
Clinical Benefit Rate (CBR) | Tumor assessments every 6 weeks from Baseline until radiographical progressive disease (PD), death (whichever occurred first), up to the primary completion date (up to 2 years)
  Clinical benefit rate was defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR) or stable disease（SD）>6 months determined by investigator using RECIST v1.1 on two consecutive occasions ≥4 weeks apart.
Number of Adverse Events using NCI CTCAE 5.0 [Safety and Tolerability] | From signing the informed consent to 30 days after last dose
  Number of Adverse Events using NCI CTCAE 5.0
Overall survival（OS） | From date of the patient starts treatment of inetetamab combined with pyrotinib and vinorelbine and vinorelbine and death from any cause，assessed up to about 48 months.
  Overall survival (OS) is defined as the time from the date of first dosing till death due to any cause.
Duration of Respons（DoR） | Tumor assessments every 6 weeks from Baseline until radiographical progressive disease (PD), death (whichever occurred first), up to the primary completion date (up to 2 years)
  The duration of respons refers to the time from the first assessment of CR or PR to the first assessment of PD or (for any reason) death, that is, the time during which the tumor continues to shrink after the patient receives a certain treatment plan.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat sen Memorial Hospital of Sun Yat sen University Shenzhen Shantou Central Hospital, Shanwei, Guangdong, China